CLINICAL TRIAL: NCT05215353
Title: Music Therapy vs. Cognitive-Behavioral Therapy for Cancer-related Anxiety (MELODY)
Brief Title: A Study Comparing Music Therapy and Cognitive Behavioral Therapy for Anxiety in Cancer Survivors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-516
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Survivorship
Keywords: Music Therapy; Cognitive Behavioral Therapy; Anxiety; 21-516
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The proposed MELODY trial is a two-arm, parallel group, randomized clinical trial (RCT) to compare the effectiveness of music therapy (M) versus cognitive behavioral therapy (CBT) for anxiety and co-morbid symptoms in a diverse, heterogeneous sample of 300 cancer survivors.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Therapy (MT) (Experimental): MT is a non-pharmacological, evidence-based intervention, in which board-certified music therapists engage patients in personally tailored experiences with music to achieve therapeutic goals. Patients will receive a workbook with materials for each session These experiences range from music-guided relaxation to more active forms of musical engagement, including singing and improvising music.
  Interventions: Other: Music Therapy; Other: assessments
- Cognitive Behavioral Therapy (CBT) (Active Comparator): Cognitive behavioral therapy (CBT) is an evidence-based, nonpharmacological intervention delivered by licensed mental health providers. Informed by the cognitive behavior model of anxiety, CBT focuses on the relationship between thoughts, behaviors, and emotions and how thoughts and behaviors can exacerbate or reduce anxiety.
  Interventions: Other: Cognitive Behavioral Therapy; Other: assessments
- Sub-study for N=18 cancer survivors original MELODY protocol for group delivery (non randomized) (Experimental): Participants will attend seven weekly 60-minute virtual group sessions, delivered through Zoom's HIPAA-compliant, encrypted, passcode-protected videoconferencing platform.
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — Participants will receive seven weekly 60-minute treatments of music therapy. All sessions will be delivered virtually through Zoom.
  Arms: Music Therapy (MT); Sub-study for N=18 cancer survivors original MELODY protocol for group delivery (non randomized)
Other: Cognitive Behavioral Therapy — Participants will receive seven weekly 60-minute treatment of cognitive behavioral therapy. All sessions will be delivered virtually through Zoom.
  Arms: Cognitive Behavioral Therapy (CBT)
Other: assessments — Participants will complete study assessments prior to randomization (week 0) and at weeks 4, 8, 16, and 26. A subgroup of 60 survivors will complete optional semi-structured interviews after treatment to understand their unique experiences with MT or CBT. All participants will be followed for 26 weeks.
  Arms: Cognitive Behavioral Therapy (CBT); Music Therapy (MT)

SUMMARY:
The researchers are doing this study to compare how music therapy and cognitive behavioral therapy, given virtually, may be able to reduce anxiety in people who have had cancer. In addition, this study will see if certain factors affect how well participants respond to music therapy or cognitive behavioral therapy. For example, the researchers will see if personal characteristics (like age, sex, race, and education) and ways of thinking (like expectations of therapy) may affect how well participants respond.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* 18 years or older
* Prior cancer diagnosis of any type or stage
* Free of oncological disease, or stable disease with no evidence of progression
* Score of ≥8 on the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
* Report anxiety symptoms lasting at least one month
* Willing to adhere to all study-related procedures, including randomization to one of two treatment arms: MT or CBT
* Access to Zoom and a quiet/private location

Inclusion Criteria for Advanced Cancer Sub-Study (N=50)

* English-speaking
* 18 years or older
* Advanced cancer diagnosis: stage III or IV lung cancer; any stage pancreatic cancer, unresectable cholangiocarcinoma, unresectable liver cancer, unresectable ampullary or peri-ampullary cancer, or other stage IV gastrointestinal cancer; stage III or IV ovarian or fallopian tube cancers or other stage IV gynecologic cancer; stage IV breast cancer; stage III testicular cancer or any stage IV genitourinary cancer; stage IV sarcoma; stage IV melanoma; stage IV endocrine cancer; lymphoma, myeloma, or leukemia
* Currently receiving oncological treatment or on active surveillance
* Karnofsky performance score of ≥60
* Score of ≥8 on the HADS anxiety subscale
* Anxiety symptoms lasting for at least 1 month
* Greater than 6-month expected survival as judged by the treating oncologist
* Willing to adhere to all study procedures
* Access to Zoom and a quiet/private location

Inclusion Criteria for group MT sub-study (N=18)

* English-speaking
* 18 years or older
* Prior cancer diagnosis of any type or stage
* Free of oncological disease, or stable disease with no evidence of progression
* Score of ≥8 on the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
* Report anxiety symptoms lasting at least one month
* Willing to adhere to all study-related procedures
* Access to Zoom and a quiet/private location

Exclusion Criteria:

* Completed active cancer treatment (e.g., surgery, radiation, chemotherapy) less than one month prior to enrollment (maintenance hormonal or targeted therapies are allowed).
* Active suicidal ideation, bipolar disorder, schizophrenia, or substance abuse
* Score of ≥10 indicative of cognitive impairment on the Blessed Orientation-Memory-Concentration
* Received a treatment course of seven or greater MT or CBT sessions for anxiety symptoms within the last six months
* Unable to provide informed consent for themselves

Exclusion Criteria for Advanced Cancer Sub-Study

* Active suicidal ideation; bipolar disorder, schizophrenia, or substance abuse
* Score of ≥10 on Blessed Orientation-Memory-Concentration
* Prior receipt of MT within the past six months
* Plan to receive any form of psychotherapy in the coming 8 weeks
* Initiation or change in anxiety medications within the past 4 weeks
* Plan to initiate or change anxiety medications in the coming 8 weeks
* Unable to provide informed consent for themselves

Exclusion Criteria for group MT sub-study

* Completed active cancer treatment (e.g., surgery, radiation, chemotherapy) less than one month prior to enrollment (maintenance hormonal or targeted therapies are allowed).
* Active suicidal ideation; bipolar disorder, schizophrenia, or substance abuse
* Score of ≥10 on Blessed Orientation-Memory-Concentration
* Prior receipt of MT within the past six months
* Plan to receive any form of psychotherapy in the coming 8 weeks
* Initiation or change in anxiety medications within the past 4 weeks
* Unable to provide informed consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
HADS anxiety score changes | 8 weeks
  Using the seven-item anxiety sub-scale of the Hospital Anxiety and Depression Scale (HADS). A score of ≥8 indicates presence of anxiety symptoms.
HADS anxiety score changes | 26 weeks
  Using the seven-item anxiety sub-scale of the Hospital Anxiety and Depression Scale (HADS). A score of ≥8 indicates presence of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- [Derived] Liou KT, Bradt J, Currier MB, Baser R, Panageas K, MacLeod J, Walker D, Li SQ, Lopez AM, McConnell K, Mao JJ. Music Therapy Versus Cognitive Behavioral Therapy via Telehealth for Anxiety in Survivors of Cancer: A Randomized Clinical Trial. J Clin Oncol. 2026 Feb 10;44(5):375-385. doi: 10.1200/JCO-25-00726. Epub 2026 Jan 6. PMID 41494146
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm